CLINICAL TRIAL: NCT05721989
Title: A Comparative Bioavailability Study of a Single Dose of Ziltivekimab Formulation B in a Manual Syringe, Formulation D in a Manual Syringe and Formulation C in a Pen-injector
Brief Title: A Research Study Looking Into Blood Levels of Three Different Formulations of the Study Medicine Ziltivekimab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN6018-4951; 2022-001862-37 (EudraCT Number); U1111-1277-3676 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ziltivekimab B (manual syringe) (Experimental): Participants will receive a single subcutaneous (s.c.) injection of 15 milligram (mg) ziltivekimab B (15 milligrams per milliliter [mg/mL]) by single-use pre-filled manual syringe on Day 1.
  Interventions: Drug: Ziltivekimab B
- Ziltivekimab D (manual syringe) (Experimental): Participants will receive a single s.c. injection of 15 mg ziltivekimab D (15 mg/mL) by single-use pre-filled manual syringe on Day 1.
  Interventions: Drug: Ziltivekimab D
- Ziltivekimab C (pen-injector) (Experimental): Participants will receive a single s.c. injection of 15 mg ziltivekimab C (30 mg/mL) by single-use pre-filled syringe assembled into a shield-activated pen-injector on Day 1.
  Interventions: Drug: Ziltivekimab C

INTERVENTIONS:
Drug: Ziltivekimab B — Participants will receive a single s.c. injection of 15 mg ziltivekimab B (15 mg/mL) by single-use pre-filled manual syringe on Day 1.
  Arms: Ziltivekimab B (manual syringe)
Drug: Ziltivekimab D — Participants will receive a single s.c. injection of 15 mg ziltivekimab D (15 mg/mL) by single-use pre-filled manual syringe on Day 1.
  Arms: Ziltivekimab D (manual syringe)
Drug: Ziltivekimab C — Participants will receive a single s.c. injection of 15 mg ziltivekimab C (30 mg/mL) by single-use pre-filled syringe assembled into a shield-activated pen-injector on Day 1.
  Arms: Ziltivekimab C (pen-injector)

SUMMARY:
A research study to investigate how quickly and to what extent different compositions of the study medicine ziltivekimab are absorbed, transported, and eliminated from the body. Ziltivekimab is not yet approved for market. The study medicine will be injected under the skin (this is called subcutaneous administration). Two different administration methods will be compared: a syringe and a pen-injector. A pen-injector is a device that is developed to make injections more easy and convenient. They are for example used by diabetes patients to inject insulin. It will also be investigated how safe ziltivekimab is and how well it is tolerated when it is used by healthy participants. Ziltivekimab has already been administered to patients with chronic kidney disease or rheumatoid arthritis. The current study will be the first study where ziltivekimab will be given to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-64 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 18.5 and 29.9 kilograms per square meter (kg/m^2) (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method.
* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, topical medication, highly effective contraceptives and occasional use of paracetamol, acetylsalicylic acid within 14 days before trial product administration.
* Clinical evidence of, or suspicion of, active infection at the discretion of the investigator.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
AUC0-inf, zilti, SD: Area under the ziltivekimab serum concentration-time curve from 0 hours and extrapolated to infinity after a single dose | From day 1 (pre-dose) to day 183 after a single dose
  Measured in day*microgram per milliliter (day*μg/mL).

SECONDARY OUTCOMES:
Cmax, zilti, SD: Maximum observed ziltivekimab serum concentration after a single dose | From day 1 (pre-dose) to day 183 after a single dose
  Measured in micrograms per milliliters (μg/mL).
AUC0-183 days, zilti, SD: Area under the ziltivekimab serum concentration-time curve from 0 hours to day 183 after a single dose | From day 1 (pre-dose) to day 183 after a single dose
  Measured in day*μg/mL.
tmax, zilti, SD: Time to maximum observed ziltivekimab serum concentration after a single dose | From day 1 (pre-dose) to day 183 after a single dose
  Measured in days.
t1/2, zilti, SD: Terminal half-life for ziltivekimab after a single dose | From day 1 (pre-dose) to day 183 after a single dose
  Measured in days.
Cl/F, zilti, SD: Apparent total serum clearance of ziltivekimab after a single dose | From day 1 (pre-dose) to day 183 after a single dose
  Measured in liters per day (L/day).
V/F, zilti, SD: Apparent volume of distribution of ziltivekimab after a single dose | From day 1 (pre-dose) to day 183 after a single dose
  Measured in liters (L).
AUC0-50 days, zilti, SD: Area under the ziltivekimab serum concentration-time curve from 0 hours to 50 days after a single dose | From day 1 (pre-dose) to day 50 after a single dose
  Measured in day*μg/mL.
Cmax, 0-50 days, zilti, SD: Maximum observed ziltivekimab serum concentration after a single dose | From day 1 (pre-dose) to day 50 after a single dose
  Measured in μg/mL.
tmax, 0-50 days, zilti, SD: Time to maximum observed ziltivekimab serum concentration after a single dose | From day 1 (pre-dose) to day 50 after a single dose
  Measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- ICON Budapest Phase I Unit, Budapest, Hungary
- ICON - location Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com